CLINICAL TRIAL: NCT05496816
Title: COVID-19 Associated Coagulopathy (CAC) in Septic Critically Ill Patients- a Retrospective Cohort Study
Brief Title: Coagulation Disturbances in COVID-19 Septic Patients
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Mirza Kovacevic, Anesthesiologist, Cantonal Hospital Zenica
Other Study IDs: CAC
Record Dates: First submitted 2022-08-07; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Coagulation Disorder; COVID 19 Associated Coagulopathy; Sepsis; Septic Shock
MeSH Terms: conditions — Hemostatic Disorders; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis
  Interventions: Diagnostic Test: CAC in septic patients
- Septic shock
  Interventions: Diagnostic Test: CAC in septic patients

INTERVENTIONS:
Diagnostic Test: CAC in septic patients — Data collected included demographic parameters, comorbidities, vasopressors requirement, laboratory findings, in-hospital mortality scoring and diagnostic colagulation scores. Demographic parameters were taken on the day of admission, all other variables were taken on the day of admission to the ICU and on the day of initiation of invasive mechanical ventilation or on the day of discharge from the ICU.
  Demographic parameters included age and sex of the patient, followed by comorbidities which was marked with Yes or No on the day of admission in the ICU. Mortality was assessed according to the qSOFA score and vasopressor requirements on the day of admission and on the day of initation of invasive mechanical ventilation or on the day of discharge. Laboratory analysis included analysis of platelets, neutrophils, lymphocytes, PCT, CRP, fibrinogen, D-dimer on the day of admission and on the day of initation of invasive mechanical ventilation or on the day of discharge.

SUMMARY:
Objective of this study was to determine the relationship between CAC and septic condition in COVID-19 critically ill patients. Data including age, sex, comorbidities, quick Sequential Organ Failure Assessment (qSOFA) score, vasopressors requirement, laboratory findings: platelets, neutrophils, lymphocytes, procalcitonin (PCT), C-reactive protein (CRP), fibrinogen, D-dimer, sepsis-induced coagulopathy (SIC) and disseminated intravascular coagulation (DIC) score were recorded on the day of admission and on the day of starting of invasive mechanical ventilation. Primary outcome was to establish CAC with sepsis; secondary outcome measure was incidence of CAC in sepsis and septic shock in COVID-19 critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* all adult critically ill patients tested positive for reverse transcriptase polymerase chain reaction (RT-PCR) of nasopharyngeal swabs to coronavirus 2 (SARS-CoV-2)
* patienets admitted to the ICU and presented with acute hypoxemic respirator failure

Exclusion Criteria:

* patients younger than 18,
* immunodeficient patients,
* patients with a history of malignancies,
* patients who developed septic state before admission,
* patients with a history of previous coagulopathy, liver and platelet disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was conducted in the COVID-19 Intensive Care Unit in the Department of Anesthesiology, Resuscitation and Intensive Care, Cantonal Hospital Zenica. Electronic data from 100 patients in 2021. were retrospectively analyzed after obtaining approval of the ethics committee of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with coagulation disorder | 1 year
  Laboratory analysis included analysis of platelets, neutrophils, lymphocytes, PCT, CRP, fibrinogen, D-dimer on the day of admission and on the day of initation of invasive mechanical ventilation or on the day of discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided